CLINICAL TRIAL: NCT06768437
Title: The Role of Epicardial Adiposity in Heart Failure With Preserved Ejection Fraction
Acronym: EAT HFpEF
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 1003
Record Dates: First submitted 2024-11-28; First posted 2025-01-10 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFPEF)
Keywords: Heart failure; Heart failure with preserved ejection fraction; Epicardial adipose tissue; Adiposity
MeSH Terms: conditions — Heart Failure; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with HFpEF: Obese and non-obese participants with heart failure with preserved ejection fraction

SUMMARY:
In this study the investigators are aiming to recruit 130 patients with heart failure with preserved ejection fraction who are obese and non-obese to undergo CT and MRI scans, as well as some other investigations including blood tests, to help investigate if having more fat around the heart leads to worse heart function in this condition. This may lead to the development of new treatments aimed at lowering fat levels around the heart and in the rest of the body, specifically to treat HFpEF.

DETAILED DESCRIPTION:
Dysregulated adipose tissue, in particular epicardial adipose tissue (EAT; fat around the heart) may be central to the pathogenesis of obesity related HFpEF. Existing studies have been limited by selection bias (only including obese cohorts), limited cardiac structural and functional assessment (primarily using echocardiography) and lack of corroborating biological data to imply causality. Pilot data demonstrate important associations between EAT with concentric LV remodelling in cohorts at high risk of HFpEF.

Further exploration of the role of EAT and other ectopic fat depots in patients with HFpEF with and without obesity, will provide novel insights into mechanisms by which adiposity drives development of HFpEF.

In this single centre, prospective, case-control study the investigators will recruit participants with HFpEF with and without obesity (total N=130) and utilise multimodality imaging to comprehensively characterise the role of excess adiposity and ectopic fat, specifically EAT, to cardiac dysfunction in HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Aged ≥18 years old
* Diagnosed with HFpEF and diagnosis confirmed by an experienced cardiologist using the HFA-PEFF diagnostic algorithm
* Echocardiogram performed within 12 months
* Able to understand written English

Exclusion Criteria:

* LV ejection fraction <45%
* Severe primary valvular heart disease
* HFpEF due to infiltrative cardiomyopathy (cardiac amyloidosis or sarcoidosis), genetic hypertrophic cardiomyopathy, restrictive cardiomyopathy/pericardial disease or congenital heart disease
* Known heritable, idiopathic or drug-induced pulmonary arterial hypertension
* Absolute contraindications to cardiac CT or MRI including estimated glomerular filtration rate (eGFR) ≤30ml/min/1.73m2. Patients with MRI-compatible devices are be excluded.
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females, aged ≥18 years old, with a diagnosis of HFpEF with and without obesity.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2037-08 (Estimated)

PRIMARY OUTCOMES:
Epicardial adipose tissue volume | At baseline
  Cardiac CT
Epicardial Adipose tissue CT attenuation | At baseline
  Cardiac CT
Left ventricular mass:volume ratio | At baseline
  Cardiac MRI

SECONDARY OUTCOMES:
Left ventricular global longitudinal strain | At baseline
  Cardiac MRI
Left ventricular circumferential peak early diastolic strain rate | At baseline
  Cardiac MRI
Myocardial blood flow | At baseline
  Cardiac MRI
left ventricular filling pressure | At baseline
  Echocardiography (Tissue Doppler)
Six minute walk test | At baseline
Coronary artery plaque volume | At baseline
  Cardiac CT angiography
Left ventricular mass | At baseline
  Cardiac MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Glenfield Hospital, University Hospitals of Leicester, Leicester, Leicestershire, United Kingdom